CLINICAL TRIAL: NCT01456351
Title: Prospective Randomised Multicenter Study for Therapy Optimization of Recurrent, Progressive Low Grade Non-Hodgkin Lymphomas and Mantle Cell Lymphomas
Brief Title: Bendamustine Plus Rituximab Versus Fludarabine Plus Rituximab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Jurgen Barth, Professor Mathias Rummel, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHL 2-2003
Record Dates: First submitted 2011-10-11; First posted 2011-10-20 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma
Keywords: Event free survival; Remission rates; Toxicity; Overall survival; Efficiency costs; Recurrent low grade
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Rituximab; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bendamustine plus Rituximab (Experimental): Bendamustine 90 mg/m² d 1+2 + Rituximab 375 mg/m² d 1 q4w
  Interventions: Drug: Bendamustine plus Rituximab
- Fludarabine plus Rituximab (Active Comparator): Fludarabine 25 mg/m² d 1-3 + Rituximab 375 mg/m² d 1 q4w
  Interventions: Drug: Fludarabine 25 mg/m² d 1-3 + Rituximab 375 mg/m² d 1 q4w

INTERVENTIONS:
Drug: Bendamustine plus Rituximab — Bendamustine 90 mg/m² d 1+2 + Rituximab 375 mg/m² d 1 q4w for maximum 6 cycles
  Arms: Bendamustine plus Rituximab
Drug: Fludarabine 25 mg/m² d 1-3 + Rituximab 375 mg/m² d 1 q4w — Fludarabine 25 mg/m² d 1-3 + Rituximab 375 mg/m² d 1 q4w for maximum 6 cycles
  Arms: Fludarabine plus Rituximab

SUMMARY:
The study addresses the question if a therapy with bendamustine plus rituximab is comparable (non inferior) with the well-tried combination of fludarabine plus rituximab with regard to event free survival (EFS) in recurrent low malignant Non-Hodgkin and mantle cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological verified CD20-positive B-Cell-Lymphomas of the following entities:
* Follicular lymphoma grade 1 and 2
* Immunocytoma and lymphoplasmocytic lymphoma
* Marginal zone lymphoma, nodal and generalised
* Mantle cell lymphoma
* lymphocytic lymphoma (CLL without leucaemic characteristics)
* non-specified/classified lymphomas of low malignancy
* Recurrent disease (remission duration minimum 3 months), independent of type or quantity of prior therapies, except of Rituximab containing regimens, or if remission duration is > 1 year after Rituximab containing regimen, or refractory to prior therapy (progression under therapy or during 3 months after completion), except refractory disease to purin analogs or Bendamustine
* Need for therapy, except mantle cell lymphomas
* Stadium II (bulky disease, 7.5 cm), II or IV
* Written informed consent
* Performance status WHO 0-2
* Histology not older than 6 months

Exclusion Criteria:

* Patients not establishing all above mentioned prerequisites
* Option of a primary, potentially curative radiation therapy
* Patients refractory to Rituximab containing regimens
* Comorbidities excluding a study conform therapy:

heart attack during the last 6 months severe, medicinal not adjustable hypertonia severe functional defects of the heart (NYHA III or IV) lung (WHO grade III or IV) liver or kidney (creatinine > 2 mg/dl, GOT + GPT or bilirubin 3 x ULN, except caused by lymphoma

* Active auto immunohemolytic anemia (AIHA)
* HIV positive patients
* Active hepatitis infection
* Severe psychiatric diseases
* No compliance or non-compliance to be expected
* Pregnant or breast feeding women
* Anamnestic malignancies or secondary malignancies, not proven
* Cured/curable by surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2003-09; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | Observation till event or death, minimum 1 year
  From date of randomization until the date of first documented progression, date of detection of a secondary malignancy or date of death from any cause, whichever came first. Minimum 1 year

SECONDARY OUTCOMES:
Remission Rates | Observation till event or death, minimum 1 year
  From date of randomization until the date of first documented progression, date of detection of a secondary malignancy or date of death from any cause, whichever came first. Minimum 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- StiL Head Office; Justus-Liebig-University, Giessen, Germany

REFERENCES:
- [Background] 58. Rummel MJ et al. Bendamustine Plus Rituximab Versus Fludarabine Plus Rituximab In Patients with Relapsed Follicular, Indolent and Mantle Cell Lymphomas - Final Results of the Randomized Phase III Study NHL 2-2003 on Behalf of the StiL (Study Group Indolent Lymphomas, Germany) Blood 2010; 116: 856
- [Background] 81. Rummel MJ et al. Bendamustine Plus Rituximab Versus Fludarabine Plus Rituximab in Patients with Relapsed Follicular, Indolent, or Mantle Cell Lymphomas - 8-Year Follow-up Results of the Randomized Phase III Study NHL 2-2003 on Behalf of the StiL (Study Group Indolent Lymphomas, Germany) Blood 2014; 124:145.
- [Background] Rummel M, Kaiser U, Balser C, Stauch M, Brugger W, Welslau M, Niederle N, Losem C, Boeck HP, Weidmann E, von Gruenhagen U, Mueller L, Sandherr M, Hahn L, Vereshchagina J, Kauff F, Blau W, Hinke A, Barth J; Study Group Indolent Lymphomas. Bendamustine plus rituximab versus fludarabine plus rituximab for patients with relapsed indolent and mantle-cell lymphomas: a multicentre, randomised, open-label, non-inferiority phase 3 trial. Lancet Oncol. 2016 Jan;17(1):57-66. doi: 10.1016/S1470-2045(15)00447-7. Epub 2015 Dec 5. PMID 26655425